CLINICAL TRIAL: NCT04380636
Title: A Phase 3 Study of Pembrolizumab (MK-3475) in Combination With Concurrent Chemoradiation Therapy Followed by Pembrolizumab With or Without Olaparib vs Concurrent Chemoradiation Therapy Followed by Durvalumab in Participants With Unresectable, Locally Advanced, Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Pembrolizumab With Concurrent Chemoradiation Therapy Followed by Pembrolizumab With or Without Olaparib in Stage III Non-Small Cell Lung Cancer (NSCLC) (MK-7339-012/KEYLYNK-012)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7339-012; MK-7339-012 (Other: MSD); KEYLYNK-012 (Other: MSD); 205352 (Registry Identifier: JAPIC-CTI); 2023-503591-25-00 (Registry Identifier: EU CT); U1111-1287-5477 (Registry Identifier: UTN); 2019-003237-41 (EudraCT Number)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death Receptor 1 (PD-1, PD1); Programmed Cell Death Receptor Ligand 1 (PD-L1, PDL1); Programmed Cell Death Receptor Ligand 2 (PD-L2, PDL2); polyadenosine 5'diphosphoribose (polyADP ribose) polymerization (PARP) inhibitor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; olaparib; Etoposide; Carboplatin; Cisplatin; Paclitaxel; Pemetrexed; durvalumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- pembrolizumab+chemoradiation→pembrolizumab+olaparib placebo (Experimental): Participants will receive pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) in combination with 3 cycles of the investigator's choice of platinum doublet chemotherapy and concurrent standard thoracic radiotherapy (60 Gray (Gy) over 6 weeks) followed by pembrolizumab plus olaparib placebo twice a day (BID) for approximately 1 year.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for olaparib; Drug: Etoposide; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed; Radiation: Thoracic Radiotherapy
- pembrolizumab+chemoradiation→pembrolizumab+olaparib (Experimental): Participants will receive pembrolizumab 200 mg IV Q3W in combination with 3 cycles of the investigator's choice of platinum doublet chemotherapy and concurrent standard thoracic radiotherapy (60 Gy over 6 weeks) followed by pembrolizumab plus olaparib 300 mg BID for approximately 1 year.
  Interventions: Biological: Pembrolizumab; Drug: Olaparib; Drug: Etoposide; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed; Radiation: Thoracic Radiotherapy
- chemoradiation→durvalumab (Active Comparator): Participants will receive 3 cycles of the investigator's choice of platinum doublet chemotherapy with concurrent standard thoracic radiotherapy (60 Gy over 6 weeks) followed by durvalumab 10 mg/kg every 2 weeks (Q2W) for approximately 1 year.
  Interventions: Drug: Etoposide; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed; Radiation: Thoracic Radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Biological: Pembrolizumab — intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: pembrolizumab+chemoradiation→pembrolizumab+olaparib; pembrolizumab+chemoradiation→pembrolizumab+olaparib placebo
Drug: Olaparib — oral tablets
  Other Names: LYNPARZA®; MK-7339; AZD2281; KU-0059436
  Arms: pembrolizumab+chemoradiation→pembrolizumab+olaparib
Drug: Placebo for olaparib — oral tablets
  Arms: pembrolizumab+chemoradiation→pembrolizumab+olaparib placebo
Drug: Etoposide — IV infusion
  Other Names: VEPESID®
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
Drug: Cisplatin — IV infusion
  Other Names: PLATINOL®
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Pemetrexed — IV infusion
  Other Names: ALIMTA®
Radiation: Thoracic Radiotherapy — external beam radiation
Drug: Durvalumab — IV infusion
  Other Names: IMFINZI®
  Arms: chemoradiation→durvalumab

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab in combination with concurrent chemoradiation therapy followed by either pembrolizumab with olaparib placebo (Arm 1) or with olaparib (Arm 2) compared to concurrent chemoradiation therapy followed by durvalumab (Arm 3) in participants with unresectable, locally advanced NSCLC. Arms 1 and 2 will be studied in a double-blind design and Arm 3 will be open-label. The primary hypotheses are:

1. Pembrolizumab with concurrent chemoradiation therapy followed by pembrolizumab with olaparib is superior to concurrent chemoradiation therapy followed by durvalumab with respect to progression-free survival (PFS) and overall survival (OS)
2. Pembrolizumab with concurrent chemoradiation therapy followed by pembrolizumab is superior to concurrent chemoradiation therapy followed by durvalumab with respect to PFS and OS

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically (histologically or cytologically) confirmed diagnosis of NSCLC
* Has Stage IIIA, IIIB, or IIIC NSCLC by American Joint Committee on Cancer Version 8
* Is unable to undergo surgery with curative intent for Stage III NSCLC
* Has no evidence of metastatic disease indicating Stage IV NSCLC
* Has measurable disease as defined by RECIST 1.1
* Has not received prior treatment (chemotherapy, targeted therapy or radiotherapy) for Stage III NSCLC; participants who have received neoadjuvant and/or adjuvant therapy for early stage disease are not eligible
* Has provided a tumor tissue sample (tissue biopsy [core, incisional, or excisional])
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 assessed within 7 days prior to the first administration of study intervention
* Has a life expectancy of at least 6 months
* A male participant must agree to use contraception and refrain from donating sperm during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention unless confirmed to be azoospermic (vasectomized or secondary to medical cause). The length of time required to continue contraception for each study intervention is as follows: Olaparib, platinum doublet, and radiotherapy: 90 days
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and agrees to use contraception and refrain from donating eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during the treatment period and for at least the time needed to eliminate each study intervention after the last dose of study intervention and agrees to abstain from breastfeeding during the study intervention period and for at least 120 days after the last dose of study intervention. The length of time required to continue contraception for each study intervention is as follows: Pembrolizumab: 120 days; Olaparib, platinum doublet, and radiotherapy: 180 days
* Has a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours for urine or within 72 hours for serum before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Has had her medical history, menstrual history, and recent sexual activity reviewed by the investigator to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Has adequate pulmonary function tests
* Has adequate organ function
* Has provided written informed consent

Exclusion Criteria:

* Has small cell lung cancer or a mixed tumor with presence of small cell elements
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Has had documented weight loss >10% (from baseline) in the preceding 3 months
* Has received prior radiotherapy to the thorax, including radiotherapy to the esophagus, mediastinum, or for breast cancer
* Has received prior therapy with an anti-programmed cell death 1 (ant-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti- programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has received prior therapy with olaparib or with any other polyadenosine 5'diphosphoribose (polyADP ribose) polymerization (PARP) inhibitor
* Has had major surgery <4 weeks prior to the first dose of study treatment (except for placement of vascular access)
* Is expected to require any other form of antineoplastic therapy, while on study
* Has received a live or live attenuated vaccine within 30 days before the first dose of study intervention; administration of killed vaccines is allowed
* Has received colony-stimulating factors (e.g., granulocyte colony-stimulating factor [GCSF], granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study treatment
* Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (e.g. bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study
* Is currently receiving either strong (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 grams per day, for at least 2 days before, during, and for at least 2 days after administration of pemetrexed
* Is unable/unwilling to take folic acid, vitamin B12, and dexamethasone during administration of pemetrexed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study treatment
* The presence of uncontrolled, potentially reversible cardiac conditions, as judged by the investigator or has congenital long QT syndrome
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ (excluding carcinoma-in situ-of the bladder) that have undergone potentially curative therapy
* Has severe hypersensitivity (≥Grade 3) to study intervention and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has active tuberculosis (TB; Mycobacterium tuberculosis) and is receiving treatment
* Has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Is considered a poor medical risk due to a serious, uncontrolled medical disorder or nonmalignant systemic disease in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 48 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 72 months
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AE) | Up to approximately 72 months
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Discontinuation Rate of Study Intervention Due to an Adverse Event (AE) | Up to approximately 72 months
  An AE is defined as as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 72 months
  ORR is defined as the percentage of participants who have achieved a Complete Response (CR) or a Partial Response (PR).
Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 72 months
  DOR is defined as the time from first documented evidence of Complete Response (CR) or a Partial Response (PR) until disease progression or death due to any cause, whichever occurs first.
Change from Baseline in EORTC Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Scale Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 scale scores will be presented.
Change From Baseline in Cough Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module 13 (EORTC QLQ-LC13) Item 1 Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-LC13 is a supplemental lung cancer-specific questionnaire that includes a single-item scale score for cough (Item 1). For this item, individual responses to the question "How much did you cough?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-LC13 cough scale score will be presented.
Change From Baseline in Chest Pain Using the EORTC QLQ-LC13 Item 10 Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-LC13 is a supplemental lung cancer-specific questionnaire that includes a single-item scale score for chest pain (Item 10). For this item, individual responses to the question "Have you had pain in your chest?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-LC13 chest pain scale score will be presented.
Change From Baseline in Dyspnea Using the EORTC QLQ-C30 Item 8 Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients and includes a single-item scale score for dyspnea (Item 8). Participant responses to the question "Were you short of breath? are scored on a 4-point scale (1=not at all to 4=very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-C30 dyspnea scale score will be presented.
Change From Baseline in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The physical functioning scale consists of participant responses to 5 questions regarding performance of daily activities [1) strenuous activities; 2) long walks; 3) short walks; 4) bed/chair rest; and 5) needing help with eating, dressing, washing themselves or using the toilet]. Participant responses are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a higher score indicating a better quality of life. The change from baseline in the EORTC QLQ-C30 physical functioning scale score will be presented.
Change from Baseline in Role Functioning Using the EORTC QLQ-C30 Items 6-7 Score | Baseline (at randomization) and at the end of study (approximately 72 months post randomization)
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The role functioning scale consists of participant responses to 2 questions regarding limitations in doing work or other activities and pursuing hobbies or leisure activities. Participant responses are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a higher score indicating a better quality of life. The change from baseline in the EORTC QLQ-C30 role functioning scale score will be presented.
Time to Deterioration (TTD) in HRQoL Using the EORTC QLQ-C30 Items 29 and 30 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-C30 Items 29 and 30 scale scores. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
TTD in Cough Using the EORTC QLQ-LC13 Item 1 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-LC13 Item 1 scale score. The EORTC QLQ-LC13 is a supplemental lung cancer-specific questionnaire that includes a single-item scale score for cough (Item 1). For this item, individual responses to the question "How much did you cough?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome.
TTD in Chest Pain Using the EORTC QLQ-LC13 Item 10 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-LC13 Item 10 scale score. The EORTC QLQ-LC13 is a supplemental lung cancer-specific questionnaire that includes a single-item scale score for chest pain (Item 10). For this item, individual responses to the question "Have you had pain in your chest?" are given on a 4-point scale (1=Not at all; 4=Very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome.
TTD in Dyspnea Using the EORTC QLQ-C30 Item 8 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-C30 Item 8 scale score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients and includes a single-item scale score for dyspnea (Item 8). Participant responses to the question "Were you short of breath? are scored on a 4-point scale (1=not at all to 4=very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a lower score indicating a better outcome.
TTD in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-C30 Items 1-5 scale scores. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The physical functioning scale consists of participant responses to 5 questions regarding performance of daily activities [1) strenuous activities; 2) long walks; 3) short walks; 4) bed/chair rest; and 5) needing help with eating, dressing, washing themselves or using the toilet]. Participant responses are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a higher score indicating a better quality of life.
TTD in Role Functioning Using the EORTC QLQ-C30 Items 6-7 Score | Up to approximately 72 months post randomization
  TTD is defined as the time to first onset of a ≥10-point decrease from baseline for EORTC QLQ-C30 Items 6-7 scale scores. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The role functioning scale consists of participant responses to 2 questions regarding limitations in doing work or other activities and pursuing hobbies or leisure activities. Participant responses are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100, with a higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (205):
- United States (33):
  - University of South Alabama, Mitchell Cancer Institute ( Site 0003), Mobile, Alabama
  - St. Bernards Medical Center ( Site 0089), Jonesboro, Arkansas
  - St Joseph Heritage Healthcare-Oncology ( Site 0088), Fullerton, California
  - Long Beach Memorial Medical Center ( Site 0006), Long Beach, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0013), Los Angeles, California
  - St. Joseph Heritage Healthcare Local Lab ( Site 0011), Santa Rosa, California
  - Torrance Memorial Physician Network / Cancer Center ( Site 0093), Torrance, California
  - Memorial Regional Hospital-Memorial Cancer Institute ( Site 0095), Hollywood, Florida
  - Miami VA Healthcare System ( Site 0024), Miami, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0022), Orange City, Florida
  - Orlando Health, UF Health Cancer Center Inc ( Site 0092), Orlando, Florida
  - Fort Wayne Medical Oncology and Hematology ( Site 0094), Fort Wayne, Indiana
  - Parkview Research Center ( Site 0032), Fort Wayne, Indiana
  - Franciscan Health Lafayette East ( Site 0031), Lafayette, Indiana
  - University of Kentucky ( Site 0096), Lexington, Kentucky
  - Norton Brownsboro Hospital-Norton Cancer Institute - Brownsboro ( Site 0035), Louisville, Kentucky
  - Pikeville Medical Center ( Site 0036), Pikeville, Kentucky
  - Massachusetts General Hospital ( Site 0038), Boston, Massachusetts
  - Henry Ford Hospital ( Site 0045), Detroit, Michigan
  - VA St. Louis Health Care System ( Site 0047), St Louis, Missouri
  - Washington University Siteman Cancer Center ( Site 0046), St Louis, Missouri
  - CHI Health St. Francis ( Site 0053), Grand Island, Nebraska
  - Rutgers Cancer Institute of New Jersey ( Site 0054), New Brunswick, New Jersey
  - Valley Health Systems - Ridgewood Campus ( Site 0056), Paramus, New Jersey
  - Montefiore Einstein Center ( Site 0083), The Bronx, New York
  - Novant Health Presbyterian ( Site 0081), Charlotte, North Carolina
  - Duke University Medical Center ( Site 0050), Durham, North Carolina
  - Piedmont Hematology-Oncology Associates ( Site 0080), Winston-Salem, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital ( Site 0060), Cincinnati, Ohio
  - Fox Chase Cancer Center ( Site 0063), Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 0066), Sioux Falls, South Dakota
  - Veterans Affairs Puget Sound Health Care System [Seattle, WA] ( Site 0075), Seattle, Washington
  - Cancer Care Northwest ( Site 0074), Spokane Valley, Washington
- Argentina (2):
  - Clinica Adventista Belgrano-Oncology ( Site 4002), Caba., Buenos Aires
  - Instituto Médico Río Cuarto ( Site 4003), Río Cuarto, Córdoba Province
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre ( Site 0100), Halifax, Nova Scotia
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0102), Montreal, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0108), Montreal, Quebec
  - McGill University Health Center - Research Institute ( Site 0114), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0110), Québec, Quebec
- Chile (5):
  - OrlandiOncologia ( Site 0201), Providencia, Region M. de Santiago
  - Bradfordhill ( Site 0200), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0202), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0203), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 0204), Antofagasta
- China (25):
  - Peking Union Medical College Hospital ( Site 3201), Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 3213), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3212), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3224), Beijing, Beijing Municipality
  - Daping Hospital,Third Military Medical University ( Site 3235), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3226), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 3219), Xiamen, Fujian
  - Peking University Shenzhen Hospital ( Site 3216), Shenzhen, Guangdong
  - Cancer Hospital Chinese Academy Of Medical Sciences. Shenzhen Center ( Site 3200), Shenzhen, Guangdong
  - Henan Cancer Hospital ( Site 3205), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center ( Site 3222), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 3218), Wuhan, Hubei
  - Xiangya Hospital of Central South University ( Site 3637), Changsha, Hunan
  - Second Xiangya Hospital of Central-South University ( Site 3227), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3225), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3238), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 3234), Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 3206), Nanchang, Jiangxi
  - Jilin Cancer Hospital ( Site 3230), Changchun, Jilin
  - Shanghai Chest Hospital ( Site 3207), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 3220), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 3203), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 3202), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 3204), Tianjin, Tianjin Municipality
  - The 1st Affil Hosp of College of Medicine, Zhejiang Univ ( Site 3232), Hangzhou, Zhejiang
- Czechia (8):
  - Masarykuv onkologicky ustav ( Site 2206), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava ( Site 2201), Ostrava, Ostrava Mesto
  - Fakultni nemocnice Kralovske Vinohrady-Radioterapeuticka a onkologicka klinika ( Site 2200), Prague, Praha 10
  - Fakultni nemocnice v Motole ( Site 2210), Prague, Praha 5
  - Nemocnice Na Plesi s.r.o. ( Site 2202), Nová Ves pod Pleší, Pribram
  - Krajska nemocnice Liberec, a.s. ( Site 2209), Liberec
  - Vseobecna fakultni nemocnice v Praze ( Site 2208), Prague
  - Nemocnice Na Bulovce ( Site 2205), Prague
- Estonia (2):
  - North Estonia Medical Centre Foundation ( Site 1601), Tallinn, Harju
  - Tartu University Hospital ( Site 1600), Tartu, Tartu
- France (8):
  - Clinique Clairval ( Site 0802), Marseille, Bouches-du-Rhone
  - C.H.R.U. de Brest - Hopital Cavale Blanche ( Site 0806), Brest, Brittany Region
  - Centre Hospitalier Annecy Genevois ( Site 0811), Epagny Metz Tessy, Haute-Savoie
  - Clinique Teissier Groupe ( Site 0808), Valenciennes, Nord
  - Hopital Avicenne ( Site 0803), Bobigny, Seine-Saint-Denis
  - Clinique de l'Europe-Service de pneumologie ( Site 0816), Amiens, Somme
  - H.I.A. Sainte-Anne ( Site 0815), Toulon, Var
  - CHD Vendee ( Site 0807), La Roche-sur-Yon, Vendee
- Germany (9):
  - Universitätsmedizin Göttingen - Georg-August-Universität ( Site 0917), Göttingen, Lower Saxony
  - Johannes Wesling Klinikum Minden ( Site 0908), Minden, North Rhine-Westphalia
  - GEHO Muenster ( Site 0910), Münster, North Rhine-Westphalia
  - Johanna Etienne Hospital-Klinik für Onkologie ( Site 0916), Neuss, North Rhine-Westphalia
  - LungenClinic Grosshansdorf GmbH ( Site 0901), Großhansdorf, Schleswig-Holstein
  - Zentralklinik Bad Berka GmbH ( Site 0905), Bad Berka, Thuringia
  - Universitaetsklinikum Jena ( Site 0911), Jena, Thuringia
  - Charite-Universitaetsmedizin Berlin Campus Virchow-Klinikum ( Site 0900), Berlin
  - Katholisches Marienkrankenhaus gGmbH ( Site 0902), Hamburg
- Hungary (5):
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 2303), Gyula, Bekes County
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 2302), Kecskemét, Bács-Kiskun county
  - Petz Aladar Megyei Oktato Korhaz ( Site 2306), Győr, Győr-Moson-Sopron
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 2305), Budapest
  - Országos Korányi Pulmonológiai Intézet-VI. Tüdöbelosztály és Bronchológia ( Site 2309), Budapest
- Italy (8):
  - Azienda Ospedaliera Umberto I- Torrette ( Site 1009), Torrette, Ancona
  - Policlinico Agostino Gemelli ( Site 1002), Rome, Lazio
  - Istituto Clinico Humanitas Research Hospital ( Site 1000), Rozzano, Lombardy
  - Azienda Ospedaliero Universitaria Careggi ( Site 1001), Florence
  - Azienda Ospedaliera Vito Fazzi ( Site 1003), Lecce
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1008), Milan
  - Policlinico di Modena ( Site 1007), Modena
  - A.O.U. Santa Maria della Misericordia di Udine ( Site 1004), Udine
- Japan (12):
  - Kurume University Hospital ( Site 3112), Kurume, Fukuoka
  - Kobe Minimally Invasive Cancer Center ( Site 3100), Kobe, Hyōgo
  - Kanagawa Cancer Center ( Site 3101), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 3103), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3110), Takatsuki, Osaka
  - National Hospital Organization Kyushu Cancer Center ( Site 3104), Fukuoka
  - Niigata Cancer Center Hospital ( Site 3109), Niigata
  - Osaka International Cancer Institute ( Site 3106), Osaka
  - Juntendo University Hospital ( Site 3111), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 3108), Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3107), Tokyo
  - Showa Medical University Hospital ( Site 3105), Tokyo
- Latvia (2):
  - Pauls Stradins Clinical University Hospital ( Site 1501), Riga
  - Riga East Clinical University Hospital ( Site 1500), Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos-Pulmonology ( Site 4201), Kaunas, Kaunas County
  - National Cancer Institute-Department of Thoracic Surgery and Oncology ( Site 4200), Vilnius, Vilniaus Miestas
- Mexico (4):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0500), Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0508), Monterrey, Nuevo León
  - CLIMERS Clinical Medical Research ( Site 0506), Orizaba, Veracruz
  - Instituto Nacional de Cancerologia ( Site 0502), Tlalpan
- Norway (5):
  - Akershus Universitetssykehus HF ( Site 1106), Lorenskog, Akershus
  - Vestre Viken HF Drammen Sykehus ( Site 1101), Drammen, Buskerud
  - Helse Stavanger HF Stavanger Universitetssjukehus ( Site 1103), Stavanger, Rogaland
  - Oslo Universitetssykehus HF. Ulleval ( Site 1100), Oslo
  - Sykehuset Oestfold ( Site 1107), Grålum, Østfold fylke
- Peru (6):
  - Hospital Nacional Carlos Alberto Seguin Escobedo ESSALUD ( Site 0604), Arequipa, Ariqipa
  - Detecta Clínica ( Site 0607), Surquillo, Muni Metro de Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0606), Lima
  - Oncosalud ( Site 0605), Lima
  - Clinica San Gabriel ( Site 0601), Lima
  - Hospital Nacional Cayetano Heredia ( Site 0602), Lima
- Poland (4):
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2404), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 2402), Warsaw, Masovian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 2400), Gdynia, Pomeranian Voivodeship
  - SPZOZ MSWIA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie ( Site 2401), Olsztyn, Warmian-Masurian Voivodeship
- Romania (11):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 2500), Bucharest, București
  - Gral Medical SRL-Medical Oncology ( Site 2511), Bucharest, București
  - Spitalul Universitar de Urgenta Bucuresti ( Site 2508), Bucharest, București
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 2506), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 2503), Comuna Floresti, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2510), Craiova, Dolj
  - Radiology Therapeutic Center-Oncology ( Site 2502), Otopeni, Ilfov
  - S C Oncocenter Oncologie Clinica S R L-Medical Oncology ( Site 2509), Timișoara, Timiș County
  - Policlinica Oncomed SRL ( Site 2504), Timișoara, Timiș County
  - Spitalul Clinic Judetean De Urgenta Constanta ( Site 2501), Constanța
  - Institutul Regional de Oncologie Iasi ( Site 2505), Iași
- Russia (8):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 1913), Chelyabinsk, Chelyabinsk Oblast
  - MSROI named after P.A. Hertsen branch of FSBI NMRC Radiology ( Site 1903), Moscow, Moscow
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 1914), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Medical institute named after Berezin Sergey ( Site 1906), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1905), Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Oncology Hospital ( Site 1909), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 1911), Kazan', Tatarstan, Respublika
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 1910), Yaroslavl, Yaroslavl Oblast
- South Korea (9):
  - National Cancer Center ( Site 2800), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 2801), Seongnam-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 2805), Suwon, Kyonggi-do
  - Ajou University Hospital ( Site 2803), Suwon, Kyonggi-do
  - Gyeongsang National University Hospital ( Site 2804), Jinju, Kyongsangnam-do
  - Chungbuk National University Hospital ( Site 2802), Cheongju-si, North Chungcheong
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 2807), Daegu, Taegu-Kwangyokshi
  - Kangbuk Samsung Hospital ( Site 2806), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2808), Seoul
- Spain (7):
  - Hospital Universitario Puerta de Hierro (Majadahonda) ( Site 1202), Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid ( Site 1200), Pozuelo de Alarcón, Madrid
  - H.R.U Malaga - Hospital General ( Site 1206), Málaga, Malaga
  - H.U. Vall de Hebron ( Site 1201), Barcelona
  - Hospital Clinic de Barcelona ( Site 1204), Barcelona
  - Hospital Universitario Virgen Macarena ( Site 1205), Seville
  - Hospital Universitario La Fe ( Site 1203), Valencia
- Thailand (4):
  - Chulalongkorn University ( Site 3003), Bangkok, Bangkok
  - Ramathibodi Hospital. ( Site 3000), Bangkok, Bangkok
  - Chiang Mai University Maharaj Nakorn Chiang Mai Hospital ( Site 3001), Chiang Mai
  - Srinagarind Hospital. Khon Kaen University ( Site 3002), Khon Kaen
- Turkey (Türkiye) (6):
  - Ankara Bilkent Sehir Hastanesi ( Site 2002), Ankara, Adana
  - Memorial Ankara Hastanesi ( Site 2006), Ankara
  - Istanbul Uni. Cerrahpasa Tip Fakultesi ( Site 2000), Istanbul
  - Medipol Universite Hastanesi ( Site 2003), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 2001), Istanbul
  - Ege University Medical Faculty ( Site 2005), Izmir
- Ukraine (8):
  - Medical center Medikal Plaza of Ecodnipro LLC ( Site 2107), Dnipro, Dnipropetrovsk Oblast
  - SOGrigoriev Inst for Med Radiolgy and Oncology of NAMS of Ukraine-Clinical oncology and hematology ( Site 2110), Kharkiv, Kharkivs’ka Oblast’
  - Communal nonprofit enterprise "Kherson Regional Oncology Dispensary" of Kherson Regional Council ( Site 2109), Antonivka Village, Kherson Oblast
  - LLC Ukrainian Center of Tomotherapy ( Site 2105), Kropyvnytskyi, Kirovohrad Oblast
  - Medical Center of Yuriy Spizhenko LLC.-Clinical Trial ( Site 2104), Kapitanivka Village, Kyivska Oblast
  - SNPE National Cancer Institute ( Site 2101), Kyiv, Kyivska Oblast
  - Medical Center Verum ( Site 2106), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Center ( Site 2100), Kyiv
- United Kingdom (7):
  - Weston Park Hospital ( Site 1406), Sheffield, Derbyshire
  - Guys and St Thomas NHS Foundation Trust ( Site 1410), London, London, City of
  - University College Hospital NHS Foundation Trust ( Site 1403), London-Camden, London, City of
  - Royal Marsden Hospital (Sutton) ( Site 1407), London, Surrey
  - Southampton General Hospital ( Site 1400), Southampton, Worcestershire
  - Leeds Teaching Hospitals NHS Trust ( Site 1401), Leeds
  - Christie NHS Foundation Trust ( Site 1409), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Jabbour SK, Cho BC, Bria E, Kato T, Bhosle J, Gainor JF, Reguart N, Wang L, Morgensztern D, Shentu Y, Kim SJ, Souza F, Reck M. Rationale and Design of the Phase III KEYLYNK-012 Study of Pembrolizumab and Concurrent Chemoradiotherapy Followed by Pembrolizumab With or Without Olaparib for Stage III Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2022 Sep;23(6):e342-e346. doi: 10.1016/j.cllc.2022.04.003. Epub 2022 Apr 29. PMID 35618629
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26266&tenant=MT_MSD_9011